CLINICAL TRIAL: NCT03719846
Title: Continuous Sample Collection Study
Acronym: CSC
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1015
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples collected during study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will provide urine cycles from both pregnant and not pregnant volunteers to maintain the SPD sample bank.

Study volunteers, seeking to conceive will be provided with Clearblue Ovulation product to help them pinpoint their most fertile time and aid conception. All volunteers will provide daily early morning urine samples throughout the study period and keep a study diary of menses and pregnancy test results for 1 menstrual cycle.

Urine samples will be received in the clinical laboratory and aliquoted into 2.25ml amounts at stored at -80˚C until required.

The study will also gather optional information from volunteers regarding a woman's general health and stress levels when trying to conceive. This will be used to study the relationship between general health, stress and conception.

DETAILED DESCRIPTION:
This study will provide urine cycles from both pregnant and not pregnant volunteers to maintain the SPD sample bank.

Study volunteers, seeking to conceive will be recruited to the study after providing written informed consent. All volunteers will be provided with Clearblue Ovulation product to help them pinpoint their most fertile time and aid conception and be required to collect daily early morning urine samples throughout the study until pregnancy is conformed or their next menstrual period starts. Volunteers will be required to keep a daily diary of menses, sample collection and pregnancy test results. The study will last for 1 menstrual cycle.

Urine samples will be received in the clinical laboratory will be tested for the presence of hormones related to pregnancy and fertility, then aliquoted into 2.25ml amounts at stored in the SPD BioBank at -80˚C until required for product development or evaluation .

The study will also gather optional information from volunteers regarding a woman's general health and stress levels when trying to conceive. This will be used to study the relationship between general health, stress and conception.

Demographic data will be summarised. No statistical analysis will be conducted on the data.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-40 years actively trying to conceive
* At least 2 regular consecutive cycles since last pregnancy/miscarriage/or since stopping breastfeeding
* Willing to disclose their pregnancy status and provide urine samples.
* Willing to give informed consent and comply with the investigational procedures.

Exclusion Criteria:

* Conditions that contraindicated pregnancy
* Taking medication, or has known condition which means they should not get pregnant.
* Currently pregnant or breastfeeding
* Abnormal liver or kidney function
* Taking antibiotics containing tetracycline.
* Previously participated in this study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 558 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Collection of urine samples during conception cycle | 2 years
  Daily during samples collected throughout the cycle in which conception occurs

CONTACTS AND LOCATIONS:
Overall Officials: sarah Johnson, Study Director — SPD Development company Ltd.
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom